CLINICAL TRIAL: NCT01915030
Title: Protect The Impact of a High Protein Diet on the Preservation of Muscle Mass During Caloric Restriction in Middle Age and Elderly People
Brief Title: Protect - The Impact of a High Protein Diet on Preservation of Muscle Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Maastricht University (Other); Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WM002-wp3
Record Dates: First submitted 2012-07-31; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Obesity
Keywords: Muscle; Physical performance; Protein; Diet; Caloric restriction
MeSH Terms: conditions — Obesity | interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High protein diet (Experimental): High protein diet during caloric restriction
  Interventions: Other: High protein diet
- Standard protein diet (Placebo Comparator): Standard protein diet during caloric restriction
  Interventions: Other: standard protein diet

INTERVENTIONS:
Other: High protein diet — controlled feeding trail. Both arms are caloric restricted
  Arms: High protein diet
Other: standard protein diet
  Arms: Standard protein diet

SUMMARY:
The present study is designed to investigate whether a high protein diet will preserve muscle mass during caloric restriction in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese subjects (BMI 27-40 kg/m2)
* Waist circumference male:≥ 102 cm, female: ≥ 88 cm
* Willingness and ability to comply with the protocol

Exclusion Criteria:

* Renal insufficiency
* Co-morbidities
* Type 1 & 2 diabetics (Fasting glucose level ≥ 7 mmol/L)
* Cancer
* COPD
* Participation in weight loss program 3 months before the intervention
* Participation of any heavy resistance-type exercise training (>1 wk) the last 2 y.
* Intentional or unintentional weight loss (> 3 kg in the last 3 months)
* Severe loss appetite
* Diagnosed allergy to milk products
* Gastric bypass
* Supplements or medication use for weight loss
* Participation in any other intervention trial
* Women can only participate if they are postmenopausal (last period ≥ a year ago)

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Body composition | baseline and 12 weeks
  DEXA scan

SECONDARY OUTCOMES:
Physical performance | baseline and 12 weeks
  1. Short Physical Performance Battery (SPPB), maximum score is 12.
  2. Leg strength by 1 Repetition Maximum, both leg extension and leg press
  3. Handgrip strength
  4. Time to walk 400m
Blood related parameters | baseline and 12 weeks
  Glucose, insulin, HbA1c, lipid profile
Muscle related parameters | baseline and 12 weeks
  muscle biopsies (muscle fiber type)
Physical activity | baseline and 12 weeks
  Questionnaire LAPAQ - Activities of Daily Living

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, professor, Principal Investigator — Prof. Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands